CLINICAL TRIAL: NCT00709163
Title: Nesiritide as an Adjunctive Therapy for Children With Dilated Cardiomyopathy Admitted to the Intensive Care Unit
Brief Title: Nesiritide - Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Juan Alejos, MD - Principal Investigator, Department of Pediatrics, University of California Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A026
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-06

CONDITIONS: Dilated Cardiomyopathy
Keywords: Pediatric; Dilated Cardiomyopathy; Nesiritide
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Natriuretic Peptide, Brain; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Nesiritide
- 2 (Placebo Comparator)
  Interventions: Drug: 5% Dextrose

INTERVENTIONS:
Drug: Nesiritide — The patient will be given an initial bolus of 1mcg/kg and then placed on a continuous infusion of 0.01mcg/kg/min. Three hours after the start of the infusion the patient will be rebolused with 1mcg/kg and increase the continuous infusion to 0.015mcg/kg/min. This will occur again at 6 hours after the start with an increase in the continuous infusion rate to 0.02mcg/kg/min. Patients will continue on the study drug for a total of 24 hours.
  Other Names: Natrecor
  Arms: 1
Drug: 5% Dextrose — The patient will be given an initial bolus of 1mcg/kg and then placed on a continuous infusion of 0.01mcg/kg/min. Three hours after the start of the infusion the patient will be rebolused with 1mcg/kg and increase the continuous infusion to 0.015mcg/kg/min. This will occur again at 6 hours after the start with an increase in the continuous infusion rate to 0.02mcg/kg/min. Patients will continue on the study drug for a total of 24 hours.
  Arms: 2

SUMMARY:
Nesiritide is a rapid vasodilator that mimics the action of an endogenous hormone - human B-type natriuretic peptide (BNP). BNP is produced naturally in the ventricles of the heart in response to stretch.

Nesiritide decreases systemic vascular resistance (SVR), pulmonary capillary wedge pressure (PCWP), right atrial pressure (RAP), and mean pulmonary arterial pressure. Nesiritide does not affect the heart rate, but does increase the stroke volume and consequently cardiac output, resulting in a decrease in the symptoms of decompensated heart failure. It is generally well tolerated, with the major negative side effect being hypotension. When compared to standard therapy consisting of dobutamine and nitroglycerin, nesiritide had similar vasodilatory effects, but showed a lower incidence of arrhythmia.

Nesiritide has been approved for IV treatment of patients with acutely decompensated congestive heart failure. Although studies have tested the effectiveness and safety of nesiritide in adult CHF patients, this has not been done in children.

Subjects enrolled in this study will be pediatric (<21 years) patients carrying a diagnosis of dilated cardiomyopathy with decompensated congestive heart failure. The standard of care for these patients is to undergo cardiac catheterization with placement of a Swan-Ganz catheter for hemodynamic monitoring. Subjects will be randomly assigned to receive either Nesiritide or placebo (5% Dextrose). The infusion will then be continued for a total of twenty-four hours. During this one day period, measurements of systemic blood pressure, central venous pressure (right atrial pressure), pulmonary capillary wedge pressure, cardiac output, mixed venous saturation, pulmonary vascular resistance, and systemic vascular resistance will be measured at regularly scheduled intervals. The Swan-Ganz catheter will remain in place for 2 hours after the discontinuation of study drug, and then removed.

The objectives of this study are:

1. To assess the efficacy of Nesiritide therapy in decreasing the pulmonary capillary wedge pressure, right atrial pressure, and systemic vascular resistance in children with dilated cardiomyopathy.
2. To assess the efficacy of Nesiritide in decreasing pulmonary edema and increasing cardiac index in the above mentioned population.
3. To assess the safety of both bolus administration and continuous infusion of Nesiritide in children with dilated cardiomyopathy.
4. To assess the pharmacokinetics of Nesiritide in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of dilated cardiomyopathy
2. Less than 21 years of age
3. Patient admitted to the intensive care unit
4. Patient requiring placement of a Swan-Ganz catheter
5. Patient's hemodynamics or clinical condition requires the use of a Swan-Ganz catheter for 26 hours following the cardiac catheterization.
6. Patient has signed an IRB approved consent form.

Exclusion Criteria:

1. Severe hemodynamic instability including patients requiring ECMO
2. Cardiac catheterization not indicated

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mattel Children's Hospital at UCLA, Los Angeles, California, United States